CLINICAL TRIAL: NCT06842654
Title: Measurement Strategies for Assessment of Health-related Quality of Life Outcomes in Cancer Patients With Progressive Disease
Brief Title: EORTC Quality of Life Measurement Strategies in Progressive Cancer
Status: Recruiting | Type: Observational
Sponsor: University of Leeds (Other)
Responsible Party: Principal Investigator, Galina Velikova, Professor Galina Velikova, University of Leeds
Other Study IDs: IRAS333361
Record Dates: First submitted 2025-02-18; First posted 2025-02-24 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-07

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Rationale: Health-related quality of life (HRQOL) in people diagnosed with cancer is of increasing interest as an endpoint in clinical care and research. It helps keep track of patients' functioning and wellbeing, and informs the net clinical benefit of treatment. However, gathering HRQOL information becomes increasingly harder when patients experience disease progression. Therefore we need to develop measurement strategies of HRQOL within the progressive disease setting. Objective: The overall aim of the project is to develop recommendations to optimise the measurement and analysis of HRQOL outcomes of cancer patients within the progressive disease setting. The aim of this sub-study is to identify the preferences of patients, their carers as proxies, and health-care professionals (HCPs) about the research objectives, how often and how we should assess HRQOL, and how we might limit dropout over time.

Sub-study design: An international, multi-centre study using semi-structured interviews.

Procedures: Across Europe, we aim to interview adult people diagnosed with cancer who experience progressive disease (N=30), their carers as proxies (N=30), and HCPs involved in cancer care and/or research (N=15). The UK site will aim to recruit a maximum of 10 patients and 10 proxies. Patients and carers will be interviewed twice to evaluate whether preferences change over time. Study outcomes: Findings can help in optimising the measurement and analysis of HRQOL outcomes of cancer patients in the progressive disease setting. This will help to better inform both clinical decision-making and regulatory processes.

ELIGIBILITY:
Inclusion Criteria:

PATIENT- Adult (> 18 years of age)

* Histologically proven or radiologically diagnosed cancer
* Clinical and/or radiological progressive disease according to RECIST criteria
* Poor prognosis, i.e. expected survival time <3 years according to the treating physician PROXIES - Adult (> 18 years of age)
* Partner, relative or close friend of a patient who is eligible according to the criteria specified above

Exclusion Criteria:

* Participants without understanding of the official language of the country in which they live
* Participants with any psychiatric condition or cognitive impairment, as determined by the treating physician, that would hamper providing informed consent for research participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult (> 18 years of age) attending ST James University Hospital in Leeds
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-08-13 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Optimise the measurement and analysis of HRQOL outcomes | 3 months
  Interview adult people diagnosed with cancer who experience progressive disease (N=10) and their carers as proxies (N=10). Patients and carers will be interviewed twice to evaluate if preferences change over time. This will develop recommendations to optimise the measurement and analysis of HRQOL outcomes of cancer patients within the progressive disease setting.

CONTACTS AND LOCATIONS:
Locations (1):
- St James Hospital, Leeds, United Kingdom